CLINICAL TRIAL: NCT03121300
Title: Functional Outcomes for Stereotactic Body Radiotherapy of Lung Lesions in High Risk Patients
Brief Title: Functional Imaging in Lung SBRT
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: UMCC 2015.146
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Patients will have 20 mL of blood collected by venipuncture at the specified time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Risk Lung Cancer Patients
  Interventions: Other: CT Scan; Other: Lung CT; Other: MRI; Other: Walk Test; Other: SGRQ; Other: Biological Sample Collection; Other: Toxicity; Other: Cardiac Assessment

INTERVENTIONS:
Other: CT Scan — Quantitative lung SPECT-CT
Other: Lung CT — CT lung ventilation
Other: MRI — DCE MRI
Other: Walk Test — 6 minute hall walk test
Other: SGRQ — St. George Respiratory Questionnaire
Other: Biological Sample Collection — Blood Draw
Other: Toxicity — Toxicity Evaluation
Other: Cardiac Assessment — Cardiac MRI Scan

SUMMARY:
Little is known about the safety of body radiation therapy (SBRT), especially the impact on pulmonary function, quality of life, and on functional changes within the lung itself. Radiation dose constraints and capturing functional changes on imaging are not well studied in this setting.

The current study aims to evaluate the utility of advanced imaging to measure lung function prior to and after treatment and to assess the feasibility of using this data to adapt SBRT planning.

DETAILED DESCRIPTION:
Stereotactic body radiation therapy (SBRT) is becoming a new standard for unresectable lung metastases and primary lung cancers.

However, it is becoming increasingly common for patients to undergo multiple courses of lung SBRT to synchronous and/or metachronous lung lesions. Further, the indications for SBRT are being expanded to patients who have very poor pulmonary function such as FEV1 < 0.5 L or DLCO < 35% predicted, who have large tumors (>3 cm), or who have centrally located lesions that abut great vessels and mainstem bronchi. Little is known about the safety of such treatments, especially the impact on pulmonary function, quality of life, and on functional changes within the lung itself. Radiation dose constraints and capturing functional changes on imaging are not well studied in this setting.

The current study aims to evaluate the utility of advanced imaging to measure lung function prior to and after treatment and to assess the feasibility of using this data to adapt SBRT planning. SPECT/CT will be used to measure ventilation and perfusion changes while. CT ventilation scans will be used to correlate functional changes observed on diagnostic SPECT/CT. Dynamic contrast enhanced MRI (DCE-MRI) will also be used to explore local vascular changes in the treated tumor. In patients whose tumors lie close to the heart, cardiac MRI will be used to investigate whether high doses of radiation per fraction are associated with changes in cardiac function. These imaging modalities may be used to potentially predict toxicity and patient response with the ultimate goal of prospectively adapt dose to individual patient and tumor characteristics. Lung function prior to and post-treatment will also be measured as a correlate of functional imaging changes. Identifying areas of the lung that are sub-functional or low-functioning may offer an opportunity to adapt stereotactic ablations that spare functional lung thereby making SBRT treatments to higher risk patients safer.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving SBRT lung treatment and who have any one of the following high risk features:
* Lung lesion > 5 cm
* DLCO < 35%
* FEV1 < 0.5 L
* Central lung tumors (defined as within 2 cm from the proximal bronchial tree)
* Tumors that abut the great vessels, trachea, spinal cord, or esophagus
* Prior lobectomy or pneumonectomy
* Prior lung radiation (SBRT or conventional definitive lung radiation)
* Patients must be 18 years of age or older

Exclusion Criteria:

* Patients who have received targeted agents or systemic potentially radiosensitizing chemotherapy within 2 weeks of lung SBRT start
* Pregnancy or lactation
* Unable to tolerate MRI without anesthesia
* Inability cooperate with the scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High Risk Lung Cancer Patients
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Longitudinal Changes in Lung Function | From baseline to 6 months post Radiation Treatment
  To characterize longitudinal changes in lung function using SPECT/CT and CT ventilation scans in "high risk" patients undergoing standard SBRT treatments.

SECONDARY OUTCOMES:
Dosimetric Predictors to Assess Changes in Toxicity | From baseline to 6 months post Radiation Treatment
  To explore radiation dosimetric predictors and correlates of SPECT-CT and CT ventilation functional imaging that predict toxicity in these patients.
Changes in SPECT-CT Correlate with Changes in CT Ventilation | From baseline to 6 months post Radiation Treatment
  To determine if early functional changes in SPECT-CT correlate with changes in CT ventilation, pulmonary function and patient reported decrements in lung function on the St. George Respiratory Questionnaire (SGRQ).
To Assess Early Vascular Changes Using DCE-MRI | From baseline to 6 months post Radiation Treatment
  To assess early vascular changes using DCE-MRI in the lung tumor treated with SBRT as a possible predictor of tumor response.

OTHER OUTCOMES:
Changes in Cardiac Function | From baseline to 6 months post Radiation Treatment
  To explore if SBRT tumors that lie within 2 cm of the heart cause any changes in cardiac function on cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No